CLINICAL TRIAL: NCT02592044
Title: Evaluation of the Effect of Aromatherapy With Lavender Essential Oil on Pain and Anxiety During Peripheral Venous Cannulation
Brief Title: Effect of Aromatherapy on Venopuncture Pain and Anxiety
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tokat Gaziosmanpasa University (Other)
Responsible Party: Principal Investigator, Tuğba Karaman, Assistant Professor, Tokat Gaziosmanpasa University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Venpuncture pain
Record Dates: First submitted 2015-10-27; First posted 2015-10-30 (Estimated); Last update posted 2016-03-21 (Estimated); Status verified 2016-03

CONDITIONS: Pain
Keywords: pain; anxiety; Catheterization, Peripheral
MeSH Terms: conditions — Pain; Anxiety Disorders | interventions — Catheterization; Aromatherapy; lavender oil

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Aromatherapy with lavender essential oil (Experimental): The 2 drops of lavender essential oil will put on 5x5 cm gauze and the patient will inhale it for 5 minutes and during peripheral venous cannulation.
  Interventions: Procedure: peripheral venous cannulation; Procedure: Aromatherapy with lavender essential oil
- Placebo (Placebo Comparator): The 2 drops water will put on 5x5 cm gauze ant the patient will inhale it for 5 minutes and during peripheral venous cannulation.
  Interventions: Procedure: peripheral venous cannulation; Procedure: Placebo

INTERVENTIONS:
Procedure: peripheral venous cannulation — The 18 gauge venous cannula will be inserted in a peripheral vein on the back of right hand of the patient.
  Other Names: cannulation
Procedure: Aromatherapy with lavender essential oil — The two drops of lavender essential oil will be dropped into the gauze and the patient will inhale it for 5 minutes and during venous cannulation.
  Other Names: lavender
  Arms: Aromatherapy with lavender essential oil
Procedure: Placebo — The two drops of water will be dropped into the gauze and the patient will inhale it for 5 minutes and during venous cannulation.
  Arms: Placebo

SUMMARY:
The effect of aromatherapy with lavender essential oil on pain and anxiety during venipuncture will be evaluated.

DETAILED DESCRIPTION:
The anxiety and pain during venipuncture may be cause to the avoidance of the medical therapy in patient as well as adult. Aromatherapy with lavender was shown that beneficial effects on chronic pain and anxiety. It's effect on acute pain and anxiety is not exactly known. In this study, the aromatherapy with the lavender will be compared with placebo to evaluate the analgesic and anxiolytic effect during peripheral venous cannulation before surgery.

ELIGIBILITY:
Inclusion Criteria:

* be scheduled for elective surgery
* be accepted to inhale lavender

Exclusion Criteria:

* age <18 years >65 years
* preoperative pain or consumption of analgesic medication
* anxiety disorders or consumption of anxiolytic medications (i.e. SSRI, benzodiazepine)
* pregnancy or breastfeeding
* asthma, chronic obstructive pulmonary disease
* poor sense of smell
* allergy to the lavender essential oil

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2015-11; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Pain Level | Within the first 5 minutes after the peripheral venous cannula insertion process
  The pain of the patients during cannulation will be measured with Visual Analog Scale from 0 to 10.

SECONDARY OUTCOMES:
Anxiety Level | Within the first 5 minutes after the peripheral venous cannula insertion process
  The anxiety of the patient during cannulation will be measured with Visual Analog Scale from 0 to 10.
Patient Satisfaction | Within the first 15 minutes after the peripheral venous cannula insertion process
  The patients' satisfaction will be measured with 5-point likert scale with 0 to 4.

CONTACTS AND LOCATIONS:
Overall Officials: Tugba Karaman, MD, Principal Investigator — Gaziosmanpasa University
Locations (1):
- Gaziosmanpasa University Medical School, Tokat Province, Turkey (Türkiye)